CLINICAL TRIAL: NCT02619136
Title: Myocardial Ischemia and Transfusion: A Pilot, Multi-centre, Open-label Randomized Controlled Trial of Two Commonly Used Transfusion Strategies in Patients With Myocardial Infarction.
Brief Title: Myocardial Ischemia and Transfusion
Acronym: MINT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Canadian Blood Services (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP-10-2016-2619
Record Dates: First submitted 2015-11-30; First posted 2015-12-02 (Estimated); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Myocardial Infarction
Keywords: Blood Transfusion
MeSH Terms: conditions — Myocardial Infarction | interventions — Blood Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restrictive Transfusion Strategy (Experimental): We will permit but not require red cell transfusions once a hemoglobin value falls below 80 g/L (required below 70 g/L) during the 30 days following randomization
  Interventions: Procedure: Transfusion
- Liberal Transfusion Strategy (Active Comparator): We will transfuse at a transfusion threshold of 100 g/L for up to 30 days after randomization.
  Interventions: Procedure: Transfusion

INTERVENTIONS:
Procedure: Transfusion — Red Blood Cell Transfusion

SUMMARY:
MINT: A pilot, multi-centre, open-label randomized controlled trial of two commonly used transfusion strategies in patients with myocardial infarction.

DETAILED DESCRIPTION:
Heart attacks are conditions where blood flow to the heart muscle is dangerously low - eventually causing heart muscle to die. Drugs improving the blood flow, and procedures such angioplasty, are the mainstay of therapies. They will only work if there is enough oxygen transported in blood. In fact, the heart may be deprived of oxygen not only because of the heart attack itself but also because of low blood counts (or anemia). Anemia, or low blood counts, may be caused by bleeding or by conditions such as cancer, kidney failure, chronic infections or conditions such as severe arthritis. A transfusion increases the delivery of oxygen to the heart muscle. However, we do not know at what level of anemia to initiate blood transfusion to prevent permanent heart damage. Indeed, having low blood counts may be harmful but blood transfusions also carries important risks including extra fluid in the lungs and heart inability to pump effectively.

In previous studies, investigators demonstrated that giving less blood is safer in most patients. But, there is little evidence in patients with heart attack. This first pilot trial aims to make sure that a large study that will answer the question is doable. The large trial aims to determine when and how much blood to give to minimize damage. In both studies, patients who have a heart attack will be divided into two groups in the hopes of preventing patients from dying. One group will receive more blood and the other group less blood. In the pilot trial, it will be evaluated if we can recruit patients with heart attack in a timely fashion. This trial will span over 12 months. If patient recruitment goes well, investigators will move ahead with the second phase of the project involving over 3500 patients. The numbers of patients who die or have another heart attack as well as if doctors follow treatment plans will be recorded. The 5-year large scale project will provide a definitive answer to the amount and optimal timing of blood transfusion.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with hemoglobin level less than 100 g/L who present with an ST-segment Elevation Myocardial Infarction (STEMI), or Non-ST-Elevation Myocardial Infarction (NSTEMI);
* Rise in cardiac biomarker values with at least one value above the 99th percentile (preferably cardiac troponin cTn )
* Presence of one of the following:

  * symptoms of ischemia;
  * new/presumed new ST segment-T wave (ST-T) changes or new left bundle branch (LBBB);
  * development of pathological Q waves;
  * imaging evidence of new loss of viable myocardium or new regional wall motion abnormality;
  * identification of an intracoronary thrombus by angiography

Exclusion Criteria:

* Patients with uncontrolled acute bleeding at the time of randomization defined as the need for uncrossed or non-type specific blood;
* Patients who decline blood transfusion;
* Patients who have a planned cardiac surgery or immediate post-cardiac surgery;Patients who have been deemed palliative by their treatment team (no commitment to aggressive on-going care);
* If known that follow-up will not be possible at 30 days;
* Previous participation in the MINT Trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3501 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Enrollment rate | Time Frame: 6 months
  Recruitment will be estimated over a 6 months period at each center
Non-adherence | 30 days
  Non-adherence will be defined as transfusing a patient allocated to the restrictive group if the hemoglobin level is greater than 80 g/L; in the liberal group, not transfusing a patient who has a hemoglobin less than 100 g/L for at least 48 hours with at least 2 consecutive values.

SECONDARY OUTCOMES:
Recurrent non-fatal myocardial infarction | 30 days
  The 3rd Universal Definition of MI will be used. Recurrent MI within 30 days of the incident MI will require: a) an increase in troponin concentration of 20% or greater from the last measured value and b) clinical symptoms or signs including i) recurrence of ST elevation ≥0.1 mV, or new pathognomonic Q waves in at least two contiguous leads; or ii) ischemic symptoms for 20 minutes or longer. Acute myocardial infarction will be adjudicated by an independent blinded committee to minimize ascertainment bias.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Hébert, MD, Principal Investigator — Centre Hospitalier de l'Universite de Montreal
Locations (4):
- Canada (4):
  - Alberta Heart Institute, Edmonton, Alberta
  - Victoria Heart Institute, Victoria, British Columbia
  - Centre Hospitalier de l'Universite de Montreal-Hotel Dieu, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836